CLINICAL TRIAL: NCT06745011
Title: Prodromal Model of Parkinson's Disease Confined to The Peripheral Nervous System
Acronym: Prompark
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-20-24; NNF230C0082689 (Other Grant/Funding Number: The Ascending Investigator, Novo Nordisk Foundation)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Polyneuropathy; Alpha-Synucleinopathy; Lewy Body Disease; Parkinson Disease (PD); Lewy Body Dementia (LBD); Multiple System Atrophy; Autonomic Failure; Cardiac Imaging; Rapid Eye Movement Sleep Behavior Disorder; REM Sleep Behavior Disorder (iRBD); REM Behavior Disorder
Keywords: Isolated Rapid Eye Movement Sleep Behavior Disorder; REM Sleep Behavior Disorder; Polyneuropathy; Idiopathic Polyneuropathy; Cardiac MIBG Scintigraphy; Prodromal Lewy Body Disease; Lewy Body Disease; Alpha-synucleinopathy
MeSH Terms: conditions — Polyneuropathies; Synucleinopathies; Lewy Body Disease; Parkinson Disease; Multiple System Atrophy; Pure Autonomic Failure; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, cerebrospinal fluid, skin, faeces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic polyneuropathy with abnormal cardiac 123I-MIBG scintigraphy: Participants diagnosed with polyneuropathy, orthostatic hypotension or non-nocturnal blood pressure dip and abnormal cardiac 123I-MIBG scintigraphy (cardiac sympathetic dysfunction)
- Idiopathic polyneuropathy with normal cardiac 123I-MIBG scintigraphy: Participants diagnosed with polyneuropathy, orthostatic hypotension or non-nocturnal blood pressure dip and normal cardiac 123I-MIBG scintigraphy

SUMMARY:
Description of a method to detect Parkinson's disease or Parkinson's-like disease at an early stage (Prodromal Parkinson's Disease) where damage is still confined to the peripheral nervous system damage. Simultaneous collection of biological material to establish a biobank for use as prognostic biomarkers for the development of Parkinson's disease and other neurodegenerative diseases in which pathological alpha-synuclein deposits accumulate.

DETAILED DESCRIPTION:
Primary aim (baseline):

To assess the prevalence of isolated REM Sleep Behavior Disorder (iRBD) or REM sleep without atonia (RSWA) in patients with idiopathic polyneuropathy with as to without abnormal cardiac 123I-metaiodobenzylguanidine (MIBG) scintigraphy (assessment of cardiac sympathetic innervation)

Secondary aim (baseline):

To assess the prevalence of Parkinson's Disease (PD), Dementia with Lewy bodies (DLB) and Multiple System Atrophy (MSA) in patients with idiopathic polyneuropathy.

Hypothesis (baseline):

iRBD is more prevalent in patients known with idiopathic polyneuropathy and abnormal sympathetic innervation of the heart (assessed by cardiac 123I-MIBG scintigraphy) as compared to normal cardiac sympathetic innervation.

Primary aim (5-follow-up):

To assess whether patients with idiopathic polyneuropathy develop RSWA, iRBD, PD, DLB or MSA over a periode of five years.

Hypothesis (5-follow-up):

Patients known with idiopathic polyneuropathy and abnormal sympathetic innervation of the heart (assessed by cardiac 123I-MIBG scintigraphy) will convert to RSWA, iRBD, PD, DLB or MSA more often than those with normal cardiac sympathetic innervation.

Methods:

Clinical evaluation in combination with questionnaires, multi-modal imaging methods and polysomnography.

(Assessment of neuropathy: Neuropathy Impairment Score - Lower Leg (NIS-LL), Utah Early Neurological Scale (UENS), Kumamoto Neurological Scale and autonomic function test including Tilt table Test, Valsalva Maneuver, Deep Breathing Test, The Quantitative sensory axon reflex test (QSART). Cognition: The Montreal Cognitive Assessment (MoCA), Trail making Test B (TMT-B). Motor function: MDS-Unified Parkinson's Disease Rating Scale part III (MDS-UPDRS-III). Multi-modal imaging: cardiac 123I-MIBG scintigraphy, PE2I-PET-CT, MR-neuromelanin. Sleep: REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ), one-night video polysomnography (PSG).)

Statistics:

The researchers expect to enroll 100 participants with idiopathic polyneuropathy and orthostatic hypotension or abnormal 24-hour blood pressure measurement (non-nocturnal blood pressure dip) who have undergone cardiac 123I-MIBG scintigraphy. Based on preliminary results, the investigators expect that 1/3 (30 participants) will have abnormal cardiac MIBG scintigraphy (cases; suggested to have prodromal PD or DLB) and 2/3 (70 participants) with normal MIBG scintigraphy (controls). The prevalence of iRBD detected by video-PSG is assumed to be 5% in participants with normal cardiac MIBG scintigraphy and 35% in participants with abnormal MIBG scintigraphy. To achieve a power of 88%, 81 participants have to be included (54 with normal and 27 with abnormal cardiac MIBG scintigraphy). Power calculation was based on Fisher's exact-test. Fisher's exact test was used because of an expected small number of participants with video PSG-detected iRBD.

Biobank:

Simultaneously collection of body tissue/fluids: skin, blood, cerebrospinal fluid and faeces. Analysis of the levels of phosphorylated tau, total-tau and amyloid beta in cerebrospinal fluid is performed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Definite polyneuropathy without known etiology (idiopathic) AND orthostatic hypotension (active stand test) OR non-nocturnal blood pressure reduction (24 hour blood pressure measurement)

Exclusion Criteria:

* Known etiology of polyneuropathy
* A diagnosis of either dementia, Parkinson's disease, Dementia with Lewy Bodies or Multiple System Atrophy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with definite polyneuropathy (confirmed by nerve conductions study) diagnosed in Jutland, Denmark and orthostatic hypotension or non-nocturnal blood pressure reduction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2031-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with REM sleep behavior disorder (RBD) | RBD-status is assessed at two time point: Baseline (at the time of enrollment) and 5-year follow-up
  RBD-status will be assessed by one-night video-polysomnography and REM Sleep Behavior Disorder Screening questionnaire (RBDSQ). Diagnosis of RBD according to American Academy of Sleep Medicine (AASM) criteria.

SECONDARY OUTCOMES:
Number of participants with Parkinson's Disease (PD) or related alpha-synucleinopathies (Dementia with Lewy bodies (DLB), Multiple System atrophy (MSA)), REM-Sleep without atonia (RSWA) | Assessed at baseline (at the time of enrollment) and at 5-year follow-up
  Diagnosis of Parkinson's Disease according to Movement Disorder Society (MDS) Clinical Diagnostic Criteria (Postuma et al., 2015) supported by dopamine transporter imaging (18F-PE2I-PET).
  Diagnosis of Dementia with Lewy bodies according to the Dementia with Lewy Bodies Consortium (Mckeith et al., 2017)
  Diagnosis of Multiple System Atrophy according to MDS Clinical Diagnostic Criteria (Whenning et al., 2022)
  REM-sleep without atonia (RSWA) is assessed by one-night video-polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Astrid J. Terkelsen, MD, DrMedSc, PhD, Professor, Principal Investigator — Department of clinical medicine, Aarhus University and Department of Neurology, Aarhus University Hospital
Locations (1):
- Institute of Clinical Medicine, Aarhus University, Aarhus, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided